CLINICAL TRIAL: NCT03352869
Title: Research of Exenatide for Management of Reproductive and Metabolic Dysfunction in Overweight/Obese PCOS Patients With Impaired Glucose Regulation
Brief Title: Research of Exenatide for Overweight/Obese PCOS Patients With IGR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: [2017]077
Record Dates: First submitted 2017-11-09; First posted 2017-11-24 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Polycystic Ovary Syndrome; Overweight and Obesity; Disorder of Glucose Regulation
Keywords: Polycystic Ovary Syndrome; Overweight and Obesity; Impaired Glucose Regulation; Exenatide; Metformin
MeSH Terms: conditions — Polycystic Ovary Syndrome; Overweight; Obesity | interventions — Exenatide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exenatide (Experimental): Drug: Byetta Generic name: Exenatide Dosage form: 5ug and 10ug Dosage: 10-20ug/day Frequency: twice a day Duration: 3 months
  Interventions: Drug: Exenatide
- Metformin (Active Comparator): Drug: Glucophage Generic name: Metformin Dosage form: 500mg Dosage: 1500-2000mg/day Frequency: 500mg three times a day/1000mg twice a day Duration: 3 months
  Interventions: Drug: Metformin
- Combination (Experimental): Drug: Byetta and Glucophage Generic name: Exenatide Dosage form: Exenatide 5ug and 10ug; Metformin 500mg Dosage: Exenatide10-20ug/day; Metformin 1500-2000mg/day Frequency: Exenatide twice a day; Metformin 500mg three times a day/1000mg twice a day Duration: 3 months
  Interventions: Drug: Exenatide; Drug: Metformin

INTERVENTIONS:
Drug: Exenatide — Use Exenatide for 3 months to treat PCOS
  Other Names: Byetta
  Arms: Combination; Exenatide
Drug: Metformin — Use Metformin for 3 months to treat PCOS
  Other Names: Glucophage
  Arms: Combination; Metformin

SUMMARY:
Compare the therapeutic effects of exenatide, metformin and their combination for 3 months on reproductive and metabolic improvements of overweight/obese PCOS patients with impaired glucose regulation.

DETAILED DESCRIPTION:
The investigators designed a randomized control trial to compare the therapeutic effects of exenatide, metformin and their combination for 3 months on reproductive and metabolic improvements of overweight/obese PCOS patients with impaired glucose regulation. The investigators plan to enroll 183 patients. Inclusion criteria: 1) Patients who have PCOS which is diagnosed according to 2003 Rotterdam criteria; 2) Overweight / obesity diagnostic criteria is based on WHO-WPR; 3) IGR diagnostic criteria is based on 1999 WHO diagnostic criteria; 4) have been treated with dietary and behavioral intervention for 3 months but are ineffective; 5) have no use of other hypoglycemic drugs before 3 months of treatment.

Patients with serious complications (cardiovascular events and recent significant liver, kidney or lung disease within 3 months); high blood pressure (>160/100mmHg); active infection; secondary diabetes; pregnancy; alcohol abuse; allergic to GLP-1 receptor agonist or metformin are excluded.

Then the investigators plan to randomly divide the 183 patients into 3 groups: exenatide group, metformin group, and combination group, with 61 samples for each group. Each group use specific treatment (showed as the group name) for 3 months. Before and after the intervention, the blood samples would be collected to detect blood glucose, insulin, lipid profile, sex hormones, blood chemistry for liver and kidney function, hsCRP etc., as well as the anthropometric measurement and image examinations. All patients discontinue after 12 weeks of treatment and only routine lifestyle intervention is performed after that. All patients receive 75 g OGTT test and insulin releasing test again 12 weeks after drug withdrawal to observe the IGR remission rate. To accurately assess the insulin secretion of islet β-cell, 13 patients would be randomly selected from MET group and from EX group respectively to receive the two-step hyperglycemic clamp before the intervention and after 12-week treatment.

The investigators will compare the data and finally identify the treatment effect of exenatide on PCOS patients.

ELIGIBILITY:
Inclusion Criteria:

1. have PCOS which is diagnosed according to 2003 Rotterdam criteria;
2. overweight / obesity diagnostic criteria is based on WHO-WPR ;
3. IGR diagnostic criteria is based on 1999 WHO diagnostic criteria;
4. have been treated with dietary and behavioral intervention for 3 months but are ineffective;
5. have no use of other hypoglycemic drugs before 3 months of treatment.

Exclusion Criteria:

* Except for serious complications (cardiovascular events and recent significant liver, kidney or lung disease within 3 months)
* high blood pressure (>160/100mmHg)
* active infection
* secondary diabetes
* pregnancy
* alcohol abuse
* allergic to GLP-1 receptor agonist or metformin

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 183 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Improvement of intravenous blood glucose from impaired glucose regulation to normal glucose regulation | up to 12 weeks
  To compare the intravenous blood glucose of three groups 12 weeks after withdrawal. All patients discontinue after 12 weeks of treatment and only routine lifestyle intervention is performed after that. All patients receive 75 g OGTT test and insulin releasing test again 12 weeks after drug withdrawal to observe the IGR remission rate. To accurately assess the insulin secretion of islet β-cell, 13 patients would be randomly selected from MET group and from EX group respectively to receive the two-step hyperglycemic clamp before the intervention and after 12-week treatment. Remission rate = Number of patients who has normal glucose tolerance 12 weeks after withdrawal / Number of patients who completed treatments × 100%

SECONDARY OUTCOMES:
Improvement of hyperandrogenism | up to 12 weeks
  To compare the free androgen index (FAI =total serum testosterone x 100 / Sex Hormone Binding Globulin) of three groups after 12-week treatment
Improvement of blood lipid | up to 12 weeks
  To compare the circulating lipid level(triglyceride, total cholesterol, HDL-C, LDL-C, etc.) of three groups after 12-week treatment
Improvement of fatty liver | up to 12 weeks
  To compare the number of fatty liver patients diagnosed by ultrasonography of three groups after 12-week treatment

CONTACTS AND LOCATIONS:
Overall Officials: Tao Tao, MD, Study Chair — RenJi Hospital Department of Endocrinology and Metabolism
Locations (1):
- Renji Hospital Department of Endocrinology and Metabolism, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kahal H, Aburima A, Ungvari T, Rigby AS, Coady AM, Vince RV, Ajjan RA, Kilpatrick ES, Naseem KM, Atkin SL. The effects of treatment with liraglutide on atherothrombotic risk in obese young women with polycystic ovary syndrome and controls. BMC Endocr Disord. 2015 Apr 2;15:14. doi: 10.1186/s12902-015-0005-6. PMID 25880805
- [Background] Elkind-Hirsch K, Marrioneaux O, Bhushan M, Vernor D, Bhushan R. Comparison of single and combined treatment with exenatide and metformin on menstrual cyclicity in overweight women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2008 Jul;93(7):2670-8. doi: 10.1210/jc.2008-0115. Epub 2008 May 6. PMID 18460557
- [Background] Kahal H, Abouda G, Rigby AS, Coady AM, Kilpatrick ES, Atkin SL. Glucagon-like peptide-1 analogue, liraglutide, improves liver fibrosis markers in obese women with polycystic ovary syndrome and nonalcoholic fatty liver disease. Clin Endocrinol (Oxf). 2014 Oct;81(4):523-8. doi: 10.1111/cen.12369. Epub 2013 Dec 12. PMID 24256515
- [Background] Jensterle M, Kocjan T, Kravos NA, Pfeifer M, Janez A. Short-term intervention with liraglutide improved eating behavior in obese women with polycystic ovary syndrome. Endocr Res. 2015;40(3):133-8. doi: 10.3109/07435800.2014.966385. Epub 2014 Oct 20. PMID 25330463
- [Background] Jensterle Sever M, Kocjan T, Pfeifer M, Kravos NA, Janez A. Short-term combined treatment with liraglutide and metformin leads to significant weight loss in obese women with polycystic ovary syndrome and previous poor response to metformin. Eur J Endocrinol. 2014 Feb 7;170(3):451-9. doi: 10.1530/EJE-13-0797. Print 2014 Mar. PMID 24362411
- [Background] Vitek W, Alur S, Hoeger KM. Off-label drug use in the treatment of polycystic ovary syndrome. Fertil Steril. 2015 Mar;103(3):605-11. doi: 10.1016/j.fertnstert.2015.01.019. PMID 25726702
- [Result] Jensterle M, Kravos NA, Goricar K, Janez A. Short-term effectiveness of low dose liraglutide in combination with metformin versus high dose liraglutide alone in treatment of obese PCOS: randomized trial. BMC Endocr Disord. 2017 Jan 31;17(1):5. doi: 10.1186/s12902-017-0155-9. PMID 28143456
- [Derived] Tao T, Zhang Y, Zhu YC, Fu JR, Wang YY, Cai J, Ma JY, Xu Y, Gao YN, Sun Y, Fan W, Liu W. Exenatide, Metformin, or Both for Prediabetes in PCOS: A Randomized, Open-label, Parallel-group Controlled Study. J Clin Endocrinol Metab. 2021 Mar 8;106(3):e1420-e1432. doi: 10.1210/clinem/dgaa692. PMID 32995892